CLINICAL TRIAL: NCT00575848
Title: A Trial of the Effects of Glycine Loading on Clinical Symptoms and Logical Memory in Patients With Schizophrenia
Brief Title: Study of the Effects of Glycine on Symptoms and Memory in Patients With Schizophrenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment and due to personnel change there was no viable way to quantify glycine levels through imaging
Sponsor: North Suffolk Mental Health Association (Other)
Collaborators: Mclean Hospital (Other); National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: A. Eden Evins, M.D., M.P.H., Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CORRC #1-2007
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Glycine; Magnetic Resonance Spectroscopy (MRS)
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Glycine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: Glycine
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Glycine — Subjects will consume glycine twice daily, once with breakfast and once with dinner. The medication is in liquid form. They will be instructed to refrigerate the liquid until the time that they take it. Subjects start by taking 10g per day for the first 2 days. Starting on the 3rd day, subjects take 0.2g/kg (15g for a 75kg adult) per day, and increase dosage by 0.2g/kg every two days, until they reach 0.8g/kg per day, which they take for the remainder of the 6-week period.
  Arms: 1
Dietary Supplement: Placebo — Subjects will consume placebo twice daily, once with breakfast and once with dinner. The placebo is in liquid form. They will be instructed to refrigerate the liquid until the time that they take it. Subjects start by taking 10g per day for the first 2 days. Starting on the 3rd day, subjects take 0.2g/kg (15g for a 75kg adult) per day, and increase dosage by 0.2g/kg every two days, until they reach 0.8g/kg per day, which they take for the remainder of the 6-week period.
  Arms: 2

SUMMARY:
The goal of this project is to understand whether glycine is helpful for improving some symptoms of schizophrenia such as low motivation, loss of interest, and social isolation. In addition, the investigators want to find out if glycine improves memory.

This project involves a three-and-a-half month trial of glycine or placebo. A placebo looks exactly like the study drug, but it contains no active drug. Glycine is a naturally occurring substance that is a part of some of the proteins in your body. Glycine has not been approved by the FDA (Food and Drug Administration) for the treatment of schizophrenia. However, the FDA allows it to be used in research studies.

Related Study at McLean Hospital: If you would like to participate in this study of glycine versus placebo at the Freedom Trail Clinic, the investigators will ask you if you would also like to participate in a related study at McLean Hospital. The study at McLean Hospital will look at the effects of glycine and placebo on levels of glycine in the brain. The study will use magnetic resonance spectroscopy to measure brain glycine levels. The magnetic resonance (MR) scanner looks like a large cylinder with a tube running down the center. You will be asked to lie down on your back on a foam-padded table and place your head into a special holder. The table will slide you inside the "hole" of the scanner. Soft foam rubber sponges may be placed on both sides of your head for comfort and to help keep your head from moving. Because the scanner contains a strong magnet, you will be asked to remove all metal objects from your person including, but not limited to: watches, rings, necklaces, bracelets, earrings and other body piercings, belts, loose change, wallet (with credit cards), items of clothing containing magnetic materials (for example, underwire bras, certain types of zippers), and shoes. These items will be secured in a safe place until your scan is completed. You will be able to remain in your street clothes. The investigators will ask you if study staff from McLean Hospital can contact you to tell you more about the study. You may refuse to be contacted by McLean Hospital. However, if you do not participate in the study at McLean, you are not eligible for the study here at the Freedom Trail Clinic.

DETAILED DESCRIPTION:
If you agree to participate in this study, you will be taking glycine or a placebo for 12 weeks - in two 6-week periods. These two 6-week periods are separated by a 2-week "wash-out" period where you take no study medication. During one of the 6-week periods, you will be taking glycine. During the other 6-week period, you will be taking placebo. Neither you nor the study staff will know in which order you receive the glycine or placebo. In case of an emergency, we can quickly find out which medication you have been taking.

If you agree to participate in this study, we will then meet for a "screening visit" to see if you are eligible for participation in the study. You will have an interview where you will be asked about your history of psychiatric illness. We will also ask about your previous history with smoking and use of other drugs and about your current medications. We will ask you to sign an authorization form so that we can look at your medical record. We will review your medical record for medical and psychiatric diagnoses and treatment. We will check your heart rate and blood pressure. We will take a saliva (spit) sample to check for use of street drugs such as alcohol, cocaine, amphetamines, opiates, and marijuana. If you test positive for the presence of any of these substances, you will not be allowed to participate in the study. Information about drug use will not become a part of your medical record, but this information will become a part of your research record.

After you have completed this screening interview, we will arrange a date and time for you to come back for an initial assessment before the start the study. The initial assessment takes about an hour and a half. During this assessment we will ask you questions about different psychiatric symptoms that you may be having. You will be asked about your thinking, mood, unusual experiences such as hearing voices, side effects from antipsychotic medications, and smoking behavior.

You will have the carbon monoxide in your breath measured. Carbon monoxide is a gas contained in cigarette smoke, and measuring the level of carbon monoxide in your breath helps us to tell whether or not you smoke cigarettes. To measure your carbon monoxide, we will have you breathe into a small hand-held machine.

We will also ask you about your regular activities during the day and what kind of hobbies/interests you have. Then you will do a memory test where the interviewer will tell you a story and ask you to repeat it back to him.

After you have completed the initial assessment, you will begin taking the study medication. The study medication is glycine or identical placebo and is in the form of a liquid. A one-week supply of the medication will be given to you on your weekly visit to McLean Hospital. You will take one dose of medication with breakfast in the morning and the second dose of medication with dinner in the evening. You should keep the study medication refrigerated. You will take approximately 30 grams (about 1 quarter of a liter) twice per day for the first 6 weeks, but the exact amount that you will take will depend upon your weight. We will instruct you in exactly how much to take.

At the end of the first 6 weeks of the study, you will stop taking the glycine or identical placebo for 2 weeks. During the 2 weeks where you take no study medication, we will arrange for you to come in for a brief check in visit (at week 7) to ask about any side effects after you have stopped taking the medication.

After two weeks of taking no medication, you will again start taking glycine or placebo for the next 6 weeks.

You will not change your regular medications during the study. You are to continue taking all your other medications throughout the study. You should notify Dr. Evins or any of the research staff if you start to take any new medications. You will come in every week to pick up your study medications.

We ask you to come for an interview and a test of your memory four times throughout the study. The first time is the initial visit described above, before you have started taking the study medication.

The other assessments will take place 6 weeks into the study (at the end of your first 6-week period on study medication), 8 weeks into the study (after the 2-week "washout" period when you will have been taking no study medication), and 14 weeks into the study (at the end of your second 6-week period on study medication).

There will be a total of 4 blood draws that will occur on 4 separate occasions. The blood draws will take place on the same days as the scanning visits at McLean Hospital. At each blood draw, we will take about 1 tablespoon of blood. The total amount of blood we will take in the study is about 4 tablespoons.

The study will last 14 weeks. At the end of the study, you will stop taking all glycine or placebo. If you or your doctor believes that glycine has been helpful to you and you wish to take it once the study has ended, it is available through some pharmacies, and you should discuss this option with your doctor or psychiatrist.

We will ask you to attend one follow-up visit a week after the end of the study, when we will ask you about any side effects you may have experienced. We will also ask you about side effects throughout the course of the study. This follow-up visit would last about 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18-65 with DSM-IV diagnosis of schizophrenia or schizoaffective disorder by diagnostic interview and chart review
2. Clinically stable on a stable dose of antipsychotic medication (any except clozapine or olanzapine) for at least one month, no current active suicidal ideation
3. Not treated with investigational medication in the past 30 days
4. Competent to provide informed consent

Exclusion Criteria:

1. Diagnosis of dementia, neurodegenerative disease, seizure disorder, current substance abuse or dependence disorders, including alcohol, active within the last 3 months or any Axis I DSM-IV diagnosis other than schizophrenia or schizoaffective disorder
2. Serious illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease that is not stabilized such that hospitalization for treatment of that illness is likely within the next four months
3. Patients who, in the investigator's opinion, pose a current severe homicide or suicide risk
4. History of multiple head injuries with neurological sequelae or a single severe head injury with lasting neurological sequelae
5. Uncontrolled hypertension
6. Anuretic
7. Use of clozapine or olanzapine in the past month
8. Subjects who weigh more than 275 lbs
9. Subjects who are claustrophobic
10. Subjects with a history of electrolyte imbalance
11. Subjects who have lost consciousness for 30 minutes or more
12. Subjects with lifetime history of stroke
13. Subjects with myocardial infarction within the last 6 months
14. Those having a pacemaker or a heart arrhythmia
15. Source of metal in body incompatible with MRI procedures
16. Those who have ever used a dietary glycine supplement

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Scale for the Assessment of Negative Symptoms (SANS) total score | 14 weeks

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) positive symptom subscale | 14 weeks
Performance on the Logical Memory subtest of the Wechsler Memory Scale | 14 weeks
Correlations between changes in clinical symptoms and changes in brain glycine levels as measured by MRS at McLean Hospital | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: A. Eden Evins, M.D., M.P.H., Principal Investigator — Massachusetts General Hospital; Andrew Prescot, Ph.D., Principal Investigator — Mclean Hospital
Locations (2):
- United States (2):
  - Brain Imaging Center, McLean Hospital, Belmont, Massachusetts
  - Freedom Trail Clinic, Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Olney JW, Farber NB. Glutamate receptor dysfunction and schizophrenia. Arch Gen Psychiatry. 1995 Dec;52(12):998-1007. doi: 10.1001/archpsyc.1995.03950240016004. PMID 7492260
- [Background] Reveley MA, De Belleroche J, Recordati A, Hirsch SR. Increased CSF amino acids and ventricular enlargement in schizophrenia: a preliminary study. Biol Psychiatry. 1987 Apr;22(4):413-20. doi: 10.1016/0006-3223(87)90163-6. PMID 3567257
- [Background] Kurumaji A, Watanabe A, Kumashiro S, Semba J, Toru M. A postmortem study of glycine and its potential precursors in chronic schizophrenics. Neurochem Int. 1996 Sep;29(3):239-45. doi: 10.1016/0197-0186(96)00013-7. PMID 8885282
- [Background] Heresco-Levy U, Javitt DC, Ermilov M, Mordel C, Silipo G, Lichtenstein M. Efficacy of high-dose glycine in the treatment of enduring negative symptoms of schizophrenia. Arch Gen Psychiatry. 1999 Jan;56(1):29-36. doi: 10.1001/archpsyc.56.1.29. PMID 9892253
- [Background] Evins AE, Fitzgerald SM, Wine L, Rosselli R, Goff DC. Placebo-controlled trial of glycine added to clozapine in schizophrenia. Am J Psychiatry. 2000 May;157(5):826-8. doi: 10.1176/appi.ajp.157.5.826. PMID 10784481
- [Background] Prescot AP, de B Frederick B, Wang L, Brown J, Jensen JE, Kaufman MJ, Renshaw PF. In vivo detection of brain glycine with echo-time-averaged (1)H magnetic resonance spectroscopy at 4.0 T. Magn Reson Med. 2006 Mar;55(3):681-6. doi: 10.1002/mrm.20807. PMID 16453318
- [Background] Andreasen NC. The Scale for the Assessment of Negative Symptoms (SANS): conceptual and theoretical foundations. Br J Psychiatry Suppl. 1989 Nov;(7):49-58. No abstract available. PMID 2695141
- [Background] Overall, J. E. & Gorham, D. R. The brief psychiatric rating scale (BPRS). Psychol Reports 10, 799-812 (1962).
- [Background] Wechsler, D. Weschsler Adult Intelligence Scale-III (The Psychological Corporation, San Antonio, TX, 1997).
- [Background] Farber NB, Newcomer JW, Olney JW. Glycine agonists: what can they teach us about schizophrenia? Arch Gen Psychiatry. 1999 Jan;56(1):13-7. doi: 10.1001/archpsyc.56.1.13. No abstract available. PMID 9892251
- [Background] Potkin SG, Jin Y, Bunney BG, Costa J, Gulasekaram B. Effect of clozapine and adjunctive high-dose glycine in treatment-resistant schizophrenia. Am J Psychiatry. 1999 Jan;156(1):145-7. doi: 10.1176/ajp.156.1.145. PMID 9892314
- [Background] Shoham S, Javitt DC, Heresco-Levy U. Chronic high-dose glycine nutrition: effects on rat brain cell morphology. Biol Psychiatry. 2001 May 15;49(10):876-85. doi: 10.1016/s0006-3223(00)01046-5. PMID 11343684